CLINICAL TRIAL: NCT03783156
Title: Polypectomy With Hot vs Cold Snare in Small Colonic Lesions
Acronym: Polypech-c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Marina de Benito Sanz, Principal investigator, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2018-12-16; First posted 2018-12-20 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Polyp of Colon; Gastrointestinal Bleeding; Colonic Adenoma
Keywords: polypectomy snare; polypectomy complications
MeSH Terms: conditions — Colonic Polyps; Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hot snare (Other): polypectomy with hot snare
  Interventions: Procedure: hot snare
- cold snare (Other): polypectomy with cold snare
  Interventions: Procedure: cold snare

INTERVENTIONS:
Procedure: hot snare — polypectomy with hot snare
  Arms: hot snare
Procedure: cold snare — polypectomy with cold snare
  Arms: cold snare

SUMMARY:
Colonoscopy is the technique of choice for the diagnosis and prevention of colorectal cancer (CRC). The identification and extirpation of adenomas decreases the incidence of CRC by up to 76%. More than 70% of the excised lesions are less than 10 mm. There is controversy about the technique to be used (resection with cold vs hot snare) in lesions of 5-9mm. Both use a polypectomy snare. The cold snare cuts by friction, while the hot snare uses electrical current. We propose a multicenter randomized clinical trial comparing both endoscopic techniques. At least 394 injuries per group will be included, randomizing patients to whom a diagnostic colonoscopy is requested for symptoms, screening or revision protocols. Randomization will be performed stratified by center. The primary objective is the proportion of incomplete polypectomies, which will be analyzed centrally from random biopsies of the edges of the lesion. As secondary objectives, we will compare the proportion of immediate and delayed hemorrhagic complications, the evolution of postprocedural abdominal pain and the factors associated with incomplete excision in each group and the factors associated with a failed cold polypectomy. The analysis of the primary objective will be carried out by means of the z test of homogeneity without using the correction of Yates, estimating the confidence interval of the difference between both groups. The analysis will be carried out by intention to treat and per protocol.

DETAILED DESCRIPTION:
1. Introduction

   Colorectal cancer (CRC) is a major cause of morbidity and mortality worldwide. It is estimated that in 2008, 1233,000 new cases were diagnosed and more than 600,000 people died for this reason throughout the world. Colonoscopy is the technique of choice for both diagnosis and prevention, since the identification and removal of colonic adenomas reduces the incidence of CRC by up to 76%.

   Different endoscopic techniques have been developed for the removal of adenomas; The choice of some over others is made according to the size, morphology and location of the lesion.
2. Hypothesis

   Conceptual hypothesis:

   Cold snare polypectomy presents a proportion of incomplete polypectomies similar to polypectomy with hot snare.

   Operational hypothesis:

   Two endoscopic techniques will be compared from two groups created by a random assignment to one or another type of polypectomy, evaluating the proportion of non-excised polypoid tissue after it. This will be done from random biopsies of the edges of the lesion and possible macroscopic remnants
3. Objectives.

   Primary objective:

   To compare the proportion of incomplete polypectomies in both types of polypectomy (cold snare vs. hot snare).

   Secondary objectives:

   Comparing the proportion of immediate and delayed bleeding complications, total and according to the severity that they present according to the American Society of Gastroenterology (ASGE) classification.

   Comparing the evolution of abdominal pain in the 5 hours postprocedure between both groups.

   Evaluating factors associated with an incomplete extirpation in each group. Evaluating factors associated with a failed cold polypectomy.
4. Design

   Multicenter randomized clinical trial
5. Methods

Study population Patients scheduled to undergo a colonoscopy in a non-urgent setting. Patients will be invited to participate before performing the colonoscopy.

Randomization It will be done once the patient agrees to participate in the work and the first candidate polyp has been identified. Each patient will be randomized (regardless of the number of lesions per patient) so all lesions of each patient will be removed in the same way. It will be stratified by center.

Intervention Patients who meet the inclusion criteria and do not present any exclusion criteria (pre-endoscopic) will be invited to participate in the study. The informed consent will be completed according to the Spanish law 41/2002 of autonomy of the patient.

1. Endoscopic procedure The interventions will be carried out in each of the participating centers. The examinations will be performed under sedation according to the protocols established in each center. Once the first lesion is identified, the method of extirpation of the lesion will be randomized.

   * Cold Group: polypectomy with a cold snare will be carried out according to the usual standards recommended by international societies. The lesion should be placed if possible in the position equivalent to 5 o'clock on the dial, the end of the snare will be placed several millimeters from the lesion and the tip of the catheter will be angled downwards, without aspiration at any time to avoid entrapment of the submucosa.
   * Hot Group: polypectomy with snare connected to the electrosurgical unit according to the standards recommended by international societies, using a mixed current (cut-coagulation). Once the lesion is captured, the snare is pulled up to slightly separate it from the surrounding mucosa before polypectomy. Elevation of the lesion prior to polypectomy will not be performed.
   * Common evaluation: once the polypectomies are completed, the base of the polypectomies will be evaluated, taking biopsies from any suggestive area and also 2 random biopsies at the base of the polypectomy.
2. Postendoscopic follow-up After a minimum of 21 days and a maximum of 28 days from the endoscopic examination, the patient will be contacted by telephone to collect the form about the evolution of the abdominal symptoms and to collect data about the appearance of complications (questions will be asked about visits to the hospital and in a targeted manner about the most frequent symptoms of the usual complications (fever, hemorrhage, abdominal pain).
3. Histological analysis The analysis of the specimens of the polypectomies will be carried out in each center according to their usual protocol. The analysis of the biopsies of the base of the polyp will be carried out centrally by a pathologist with more than 5 years of experience in digestive pathology. Samples from the base of the polyp will be sent periodically from each center to the Salamanca university hospital through a messenger service. The pathologist will be blinded regarding the histological diagnosis of the excised polyp and the type of polypectomy (although it is true that it is difficult to blind this last point since the presence of heat artifacts in those removed with a hot handle is very frequent). The samples sent for centralized analysis will not be stored, but will be destroyed once the study is completed according to standard protocols.

Sample size Assuming a proportion of incomplete polypectomies in both groups of 10% (using the taking of biopsies as a diagnostic pattern) and setting an equivalence limit of 7%, a total of 315 lesions per group are estimated to have an α risk of 5% and a power of 80%. Assuming a proportion of losses (polyps not recovered for histological study, polypectomies of the failed Cold group of 20%), an estimated 394 lesions per group are needed, with a total of 788 lesions in total.

Data Collection All the variables concerning the characteristics of the endoscopist, the patient and the injuries included will be collected in each center. The variables related to the histological diagnosis will be collected in the same way in the respective center. The variables concerning the follow-up will be collected in a centralized manner, through a telephone call that will be made between 3 and 4 weeks from the procedure. The variable related to the histological study of the base of the polyp will be collected in a centralized manner by the pathologist in charge of the analysis of the samples.

6. Data management

Data from the data collection notebooks will be merged by the main researcher or collaborating researchers anonymously, encrypted and dissociated from the clinical information by means of a patient identification code (ID), in an online database. A copy of the database will be used in each participating center, which will be merged after completing the data collection. The responsible researcher will define an ID for each participant. The data entered in the database will be anonymous and the database will be protected with a password to which only the researchers will have access.

The unified file will be kept at the Río Hortega University Hospital and will be maintained until the end of the study. Regarding the application of the Organic Law on Data Protection 15/1999 and 1720/2007 that develops it, it should be noted that the protocol defined in the project oriented to epidemiological analysis, determines that the files will record information completely anonymized

7. Statistical analysis

The Access program (Microsoft Corporation, Edmond, USA) will be used for the realization of the database and the statistical analysis of them will be carried out through the STATA program (StataCorp, 2013. Stata Statistical Software: Release 13. College Station, StataCorp LP). In the quantitative variables, the arithmetic mean and the standard deviation will be calculated (variables that do not follow a normal distribution according to the Kolmogorov-Smirnov test will be described with median, minimum, maximum and interquartile range), and the qualitative ones will be expressed as percentages and your 95% confidence intervals.

The analysis of the primary objective, the proportion of incomplete polypectomies in both groups will be compared by means of the z test of homogeneity without using the correction of Yates.

The confidence interval of the difference between the two groups will also be estimated. The analysis will be carried out by intention to treat, regardless of the type of polypectomy performed and per protocol (assigning the lesions assigned to the group Cold that are extirpated with hot snare to the Hot group). To evaluate possible confounding factors (endoscopist, nurse, snare type, location ...), the STATA confound user command will be used, defining as a significant change that which conditions a change in the odds ratio greater than 10% with respect to the one obtained with the complete model. In case several models do not present differences greater than 10%, the most parsimonious will be chosen.

Within the secondary objectives, the proportion of complications in both groups will be verified by the de2 test. To evaluate the factors associated with incomplete polypectomies and those associated with failed cold polypectomy, multivariate logistic regression techniques will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years scheduled to undergo a colonoscopy.

Exclusion Criteria:

* Absence of lesions of 5-9 mm.
* Contraindication for polypectomy (anticoagulant treatment, treatment with clopidogrel, coagulopathy or severe thrombocytopenia)
* Loss of polypectomy specimen
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with presence of adenomatous tissue al the base of polypectomy | 3 months
  Number of patients with polypoid tissue at the base of polypectomy

SECONDARY OUTCOMES:
Number of participants with Postpolypectomy Complications | 21-28 days
  Clinical complications after polypectomy

CONTACTS AND LOCATIONS:
Overall Officials: Marina de Benito, MD, Principal Investigator — Hospital Río Hortega
Locations (1):
- Hospital Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawamura T, Takeuchi Y, Asai S, Yokota I, Akamine E, Kato M, Akamatsu T, Tada K, Komeda Y, Iwatate M, Kawakami K, Nishikawa M, Watanabe D, Yamauchi A, Fukata N, Shimatani M, Ooi M, Fujita K, Sano Y, Kashida H, Hirose S, Iwagami H, Uedo N, Teramukai S, Tanaka K. A comparison of the resection rate for cold and hot snare polypectomy for 4-9 mm colorectal polyps: a multicentre randomised controlled trial (CRESCENT study). Gut. 2018 Nov;67(11):1950-1957. doi: 10.1136/gutjnl-2017-314215. Epub 2017 Sep 28. PMID 28970290
- [Background] Noda H, Ogasawara N, Sugiyama T, Yoshimine T, Tamura Y, Izawa S, Kondo Y, Ebi M, Funaki Y, Sasaki M, Kasugai K. The Influence of Snare Size on the Utility and Safety of Cold Snare Polypectomy for the Removal of Colonic Polyps in Japanese Patients. J Clin Med Res. 2016 Sep;8(9):662-6. doi: 10.14740/jocmr2646w. Epub 2016 Jul 30. PMID 27540440
- [Background] Din S, Ball AJ, Riley SA, Kitsanta P, Johal S. A randomized comparison of cold snare polypectomy versus a suction pseudopolyp technique. Endoscopy. 2015 Nov;47(11):1005-10. doi: 10.1055/s-0034-1392533. Epub 2015 Jul 10. PMID 26165735
- [Background] Lee CK, Shim JJ, Jang JY. Cold snare polypectomy vs. Cold forceps polypectomy using double-biopsy technique for removal of diminutive colorectal polyps: a prospective randomized study. Am J Gastroenterol. 2013 Oct;108(10):1593-600. doi: 10.1038/ajg.2013.302. Epub 2013 Sep 17. PMID 24042189
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Pattullo V, Bourke MJ, Tran KL, McLeod D, Williams SJ, Bailey AA, Alexander S, Mishra A, Co J. The suction pseudopolyp technique: a novel method for the removal of small flat nonpolypoid lesions of the colon and rectum. Endoscopy. 2009 Dec;41(12):1032-7. doi: 10.1055/s-0029-1215294. Epub 2009 Nov 6. PMID 19899034
- [Background] Ichise Y, Horiuchi A, Nakayama Y, Tanaka N. Prospective randomized comparison of cold snare polypectomy and conventional polypectomy for small colorectal polyps. Digestion. 2011;84(1):78-81. doi: 10.1159/000323959. Epub 2011 Apr 14. PMID 21494037
- [Background] Aslan F, Camci M, Alper E, Akpinar Z, Arabul M, Celik M, Unsal B. Cold snare polypectomy versus hot snare polypectomy in endoscopic treatment of small polyps. Turk J Gastroenterol. 2014 Jun;25(3):279-83. doi: 10.5152/tjg.2014.5085. PMID 25141316

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT03783156/Prot_SAP_000.pdf